CLINICAL TRIAL: NCT01962649
Title: A Pilot Study of Optical Molecular Imaging for Percutaneous Biopsy of Hepatocellular Carcinoma Using Indocyanine Green
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Radiological Society of North America (Other)
Responsible Party: Principal Investigator, Umar Mahmood, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 13-314
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2018-04-25 (Actual); Status verified 2018-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Indocyanine Green

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ICG & Optical Molecular Imaging (Experimental): All patients will receive a dose of ICG 0.5mg/kg, with a maximum dose of 40mg, one day prior to the scheduled procedure. The patients will then undergo a routine image-guided biopsy on the day of the procedure; immediately prior to obtaining the biopsy sample, fluorescence intensity within the target lesion will be measured by a handheld optical molecular imaging device, which will be passed through the biopsy needle. Once the core sample is obtained using a standard biopsy needle, the specimen will be imaged using an epifluorescence, point-of-care imaging system and will then be submitted for standard pathologic analysis.
  Interventions: Biological: ICG; Device: Optical molecular imaging

INTERVENTIONS:
Biological: ICG
  Other Names: IC-Green
Device: Optical molecular imaging
  Other Names: OMI

SUMMARY:
This research study is evaluating an imaging contrast agent called indocyanine green, also known as ICG, in combination with image guided liver biopsies.

In this research study, the investigators are looking at the ability of ICG to collect within liver tumors during biopsy. The participant will be receiving a biopsy of their liver as a part of their medical care. By participating in this trial, the only additional requirement will be for the participant to come to the hospital on the day prior to their scheduled biopsy to receive an injection of ICG. During the biopsy, the investigator will measure the amount of ICG that is in the participant's liver tumor by using two experimental devices designed by the study investigators that shine light on tissue. One device consists of an imaging system attached to a small borescope that will go inside the participant's body during the biopsy. The second device shines light on the biopsy sample outside of the participant's body after the biopsy has been taken. The participant may undergo imaging with one or both of these devices.

DETAILED DESCRIPTION:
Before the research starts (screening): After signing this consent form, the participant will be asked to undergo some screening tests or procedures to find out if the participant can be in the research study. Many of these tests and procedures are likely to be part of regular care and may be done even if it turns out that the participant does not take part in the research study. If the participant has had some of these tests or procedures recently, they may or may not have to be repeated.

* A medical history, which includes questions about the participant's health, current medications, and any allergies.
* Performance status, which evaluates how the participant is able to carry on with their usual activities.
* An assessment of your liver by X-ray, ultrasound, CT (Computerized Tomography) scan, MRI (Magnetic Resonance Imaging) or PET (Positron Emission Tomography) scans.
* Anesthesia score, which evaluates how the participant tolerates the sedation given with biopsies.
* Blood tests.

If these tests show that the participant is eligible to participate in the research study, the participant will receive the study agent. If the participant does not meet the eligibility criteria, then the participant will not be able to participate in this research study.

After the screening procedures confirms that the participant is eligible to participate in the research study: The participant will be scheduled for their regular CT- or ultrasound-guided liver biopsy. On the day prior to the procedure, the participant will come to our Interventional Radiology waiting area at Massachusetts General Hospital. After the participant arrives, the participant will be interviewed by a research doctor and receive a dose of ICG intravenously. The participant will be monitored for 30 minutes after the injection, and after this time, the participant will be free to leave. On the day of the procedure, the participant will come back to the Interventional Radiology waiting area. After the participant arrives, the participant will receive an intravenous line. The participant may also have some blood drawn (no more that 4 tablespoons) for any tests needed in addition to blood work done before the participant was enrolled in the study. The participant will then meet again with the research doctor, who will go over the procedure with the participant and as usual obtain their consent to have the standard liver biopsy. The nurse will begin administering the sedatives until the participant is comfortable to proceed with the procedure. The research doctor and his assistant will advance a hollow biopsy needle through the skin and into the lesion in the liver. A miniature endoscope, small enough to fit through the hollow center of the biopsy needle, will then be passed through the needle so that the tip of the endoscope is within the lesion. The fluorescence within the lesion will be measured with the endoscope by a special camera attached to the back of the endoscope. The endoscope will then be removed, and the lesion will be biopsied with a standard biopsy needle. If the participant is undergoing a biopsy of the liver to obtain a sample of their liver tissue and not a specific area in the liver, the endoscopic imaging described above will not be performed. The biopsy will be performed in the usual way. Once the biopsy is performed, the sample of tissue from the biopsy will be imaged by a special camera and computer that will be within the procedure room. The added steps for this trial should only add approximately 5 minutes to the procedure time.

After the procedure: After the procedure is complete, the investigator will bring the participant to the recovery room so that the participant can sleep off the sedative medications. Throughout this time, the participant will be observed by a nurse, and vital signs will be monitored. The participant will be given the usual post-procedure instructions. The investigator would like to keep track of your medical condition after the procedure to make sure no side effects have occurred. The investigator would like to do this by calling the participant on the telephone the day after the procedure and 1 week after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet the following criteria on screening examination to be eligible to participate in the study:
* Participants must be patients with imaging findings revealing a focal hepatic lesion suspicious for but not diagnostic of hepatocellular carcinoma. Eligible patients will be those whose imaging demonstrates an incompletely characterized focal hepatic lesion for which either ultrasound- or CT-guided biopsy is planned.
* For the negative control study, participants must be patients without known malignancy for whom either ultrasound- or CT-guided non-focal liver biopsy is planned to evaluate a non-malignant process.
* Fit for conscious sedation for percutaneous biopsy - American Society of Anesthesiologists (ASA) Class I or II.
* Age greater than or equal to 18 years. Because no dosing or adverse event data are currently available on the use of ICG in participants <18 years of age, children are excluded from this study but will be eligible for future pediatric Phase I trials.
* Life expectancy of greater than 6 months.
* ECOG performance status <2 (see Appendix A).
* Participants must have normal organ and marrow function as defined below:
* Leukocytes > 3,000/mcL
* Absolute neutrophil count > 1,500/mcL
* Platelets > 50,000/mcL
* The effects of ICG on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who exhibit any of the following conditions at screening will not be eligible for admission into the study.
* Participants with ASA class III, IV, V.
* Participants with documented allergy to iodine or iodine containing compounds.
* Participants with documented allergy to sulfur containing compounds.
* History of adverse reactions to percutaneous procedures or sedatives for endoscopy or percutaneous biopsy.
* Participants taking phenobarbital, phenylbutazone, primidone, phenytoin, haloperidol, nitrofurantoin, and probenecid.
* Participants who are unable to discontinue warfarin and clopidogrel anticoagulation 5 days prior to the procdure.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ICG.
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study because there are unknown but potential teratogenic or abortifacient effects of ICG. Because there is an unknown but potential risk of adverse events in nursing infants secondary to treatment of the mother with ICG, breastfeeding should be discontinued if the mother is treated with ICG. These potential risks may also apply to other agents used in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2013-10 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Measurement of fluorescence intensity within focal hepatic lesions | 2 Years
  We hypothesize that HCC lesions will have significantly higher fluorescence intensity following ICG administration that normal/cirrhotic liver parenchyma. This will allow the proceduralist to recognize during the procedure whether the target lesion has been sampled accurately. We also hypothesize that OMI will characterize malignant lesions with >90% accuracy prior to core biopsy, with standard of care histology and follow up imaging as the gold standard. Benign and malignant lesions will have significantly different ICG uptake to allow for their differentiation based on their ICG fluorescence signal intensity measured percutaneously.

CONTACTS AND LOCATIONS:
Overall Officials: Umar Mahmood, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States